CLINICAL TRIAL: NCT03276455
Title: Evaluation of Safety and Efficacy of Transplantation of Autologous Hematopoietic Stem Cell Genetically Modified in Beta-Thalassemia Major
Brief Title: Gene Therapy for Beta-Thalassemia Major Using Autologous Hematopoietic Stem Cell Genetically Modified
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangdong Yike Gene Science and Technology CO.,Ltd (Industry)
Responsible Party: Principal Investigator, Chunfu Li, Director and professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NanFangHospital
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Beta Thalassemia Major
Keywords: Beta thalassemia; Gene therapy; Beta-globin; Hematopoietic stem cells; Lentiviral vector
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Beta-thalassemia major subjects who are 8 years age or older are transplated by autologous CD34+ cells genetically modified(autologous hematopoietic stem cell transduced with lentiviral vector encoding the therapeutic beta-globin gene).
  Interventions: Genetic: Autologous CD34+ cells genetically modified

INTERVENTIONS:
Genetic: Autologous CD34+ cells genetically modified — Autologous hematopoietic stem cell transduced with lentiviral vector encoding the therapeutic beta-globin gene. The target dose in the transduced product is 3x10^6 cells/Kg CD34+ cells, with a minimum dose of 2 x 10^6/Kg and a maximum dose of 20 x 10^6/Kg, depending on the yield of cells. The product will be injected intraosseously following intravenous BU ±Flu ±Cy.

SUMMARY:
This is a single group, open label study in 10 subjects who are 8 years of age or older with beta-thalassemia major. The objective of this study is to evaluate the safety and efficacy of autologous hematopoietic stem cell transduced with lentiviral vector for the treatment of beta-thalassemia major.

DETAILED DESCRIPTION:
Beta-thalassemia major is a life-threatening genetic disease of red cell malfunction. It is caused by mutations in the beta-globin gene which encodes the beta-globin protein, leading to the ineffective erythropoiesis, hemolysis and anemia. Transplantation of allogeneic hematopoietic stem cells (HSCT) is the only available cure which is, however, has the significant risk of transplant related mortality, graft versus host disease and limited source. Therefore, transplantation of autologous hematopoietic stem cells will be an attractive therapeutic treatment for beta-thalassemia major patients. 10 patients will be treated with genetically modified autologous hematopoietic stem cells which transduced with lentiviral vector encoding for beta-globin gene.

Patients will participate for this study for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 8 years of age or older.
* Subjects or their parents/legal guardians must be able to understand and voluntarily sign an informed consent form.
* Subjects must have a confirmed diagnosis of ß-thalassemia major and

  ≥100 mL/kg/year of pRBCs or ≥ 8 transfusions of pRBCs per year over a minimum of two years prior to entry onto the study.
* Subjects must be in clinically stable condition and eligible for hematopoietic stem cell transplantation.
* Subjects must satisfy Karnofsky index ≥80% for adults or Lansky index

  ≥70% for children.
* Subjects must have survival expectancy of greater than 6 months.
* Subjects must have been treated and followed up for at least the past 2 years in specialized institutions where they have comprehensive assessment of the disease（including psychiatric assessment），and detailed medical materials at least the past 2years so as to self-contrast before and after treatment.
* Subjects must discontinue treatment of hydroxyurea, 5-azoside or cytarabine at least three months prior to entry onto the study.

Exclusion Criteria:

* Having an HLA-matched donor(sibling or of a suitable 10/10 matched unrelated donor).
* Positivity for HIV (serology or RNA), and/or HbsAg and/or HBV DNA and/or HCV RNA (or negative HCV RNA but on antiviral treatment).
* Contraindication to anesthesia for bone marrow collection.
* Severe, bacterial, active viral, or fungal infection, etc.
* The history of malignant tumor.
* The white blood cell (WBC) count <3000/uL and/or platelet count <100,000/uL exclude hypersplenism factor.
* Family history of familial cancer syndromes (including but not limited to Hereditary breast and ovarian syndrome, hereditary non-polyp colorectal cancer syndrome, familial adenomatous polyposis).
* Previous allogeneic bone marrow transplantation.
* The history of psychosis and any psychiatric disorder.
* Active substance abuse, drug or alcohol abuse recently.
* The history of complex allo-immunization which could cause difficulty administering transfusions.
* Female adults who are pregnant , breast feeding or lack of effective contraception.
* History of major organ damage including:

Severe cerebrovascular disease or cognitive sequelae, including hemiplegia. Severe liver disease with alanine transaminase (ALT) >3 upper limit of normal. Severe liver cirrhosis or fibrosis on liver biopsy. Heart disease with ejection fraction<25% or T2* <10 ms by magnetic resonance imaging (MRI). Kidney disease with creatinine clearance <30% normal value. Lung disease, including pulmonary fibrosis, pulmonary arterial hypertension or pulmonary function tests below standard (i.e., pO2<90 mmHg and/or carbon dioxide diffusion coefficient<50%). Endocrine disorder including insulin dependent diabetes mellitus, Hyperthyroidism or deficiency, Hyperparathyroidism or deficiency.

* Participation in another clinical study within 30 days of screening.
* Subjects with severe iron overload determined by the researchers.
* Any other situation that unsuitably undergoing hematopoietic stem cell transplantation determined by the physicians or researchers.
* Presence of chromosomal abnormalities by bone marrow detected.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | 0-36 months after transplantation
  Evaluate the safety of treatment with transplantation of autologous hematopoietic stem cell transduced with lentiviral vector encoding the therapeutic beta-globin gene as measured by the incidence of adverse events.
hemoglobin conten | 3-36 months after transplantation
  Evaluate the efficacy of treatment with transplantation of autologous hematopoietic stem cell transduced with lentiviral vector encoding the therapeutic beta-globin gene by the detection hemoglobin content of peripheral blood cells.

SECONDARY OUTCOMES:
Hematopoietic stem cell engraftment | 42 days after transplantation
  Success and kinetics of hematopoietic stem cell engraftment.
RCL | 1-36 months after transplantation
  The generation of a replication-competent lentivirus (RCL).
VCN | 1-36 months after transplantation
  Quantify gene transfer efficiency and expression by evaluation of average vector copy number(VCN) in blood or bone marrow cells.
bete-globin content | 1-36 months after transplantation
  Evaluate the efficacy of treatment by detection of bete-globin content of HGB of peripheral blood cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospial, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No